CLINICAL TRIAL: NCT03247803
Title: Comparison of Use of a Shortened Air-Q® Self-Pressurizing Intubating Laryngeal Airway Versus the Williams Intubating Airway for Single-Operator Flexible Bronchoscopic Intubation.
Brief Title: Air-Q® SP Versus Williams Intubating Airway for Single-Operator FOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-0542
Record Dates: First submitted 2017-07-28; First posted 2017-08-14 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Intubation; Difficult or Failed; Laryngeal Masks
Keywords: Air-Q® SP; Williams Airway Intubator (WA); Flexible Bronchoscopic intubation (FBI); Fiberoptic Intubation (FOI); Fiberoptic Intubating Airway(FIA); Laryngeal Mask Airway

STUDY DESIGN:
Intervention Model Description: Adult patients presenting for a surgical or interventional procedure requiring general anesthesia and tracheal intubation, who do not meet any of the study exclusion criteria, and who give their informed consent, will be randomly allocated to receive either an air-Q SP or Williams Intubating Airway as a conduit to aid flexible bronchoscopic intubation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Each study subject will be blinded to the study device they receive; however, the anesthesia provider will not be blinded to the study device and will have access to all monitors deemed appropriate by the primary anesthesia team caring for the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air-Q SP (Experimental): air-Q Self-Pressurizing intubating Laryngeal Airway, sizes 3.5 and 4.5 (Mecury Medical, Clearwater, FL, USA)
  Interventions: Device: air-Q® SP
- Williams Intubating Airway (Experimental): Airway Intubator, Williams, Adult Female, Single Use, Molded Surlyn Plastic, 9 cm or Airway Intubator, Williams, Adult Male, Single Use, Molded Surlyn Plastic, 10 cm
  Interventions: Device: Williams Airway Intubator (WA)

INTERVENTIONS:
Device: air-Q® SP — air-Q SP placement for airway maintenance,
  Other Names: air-Q SP placement for airway maintenance
  Arms: Air-Q SP
Device: Williams Airway Intubator (WA) — WA is placed in subject's oropharynx. If the vocal cords are not in view at the end of the WA, the operator may ask an assistant to perform an airway maneuver (e.g., jaw thrust, anterior jaw lift, or lingual traction) to attempt to bring the vocal cords into view
  Other Names: WA is placed in subject's oropharynx.
  Arms: Williams Intubating Airway

SUMMARY:
The air-Q and air-Q SP are commercially-available supraglottic airways (SGAs) that can be used for primary airway maintenance or as a conduit for FOI, as can be the Williams, Ovassapian, and Berman Intubating Airways. The air-Q products have the same overall geometrical design, but differ in their cuff inflating mechanisms, where the air-Q uses a traditional pilot balloon valve, while the air-Q SP utilizes a self-inflating cuff that dynamically adjusts according to the relative resistances to airflow between the patient's lungs and the device's cuff. The purpose of this study is to compare the single-operator intubation success using the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation (FBI) and to compare the single-operator intubation success using the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation. Both devices are commercially-available and being used in the study in accordance with their labeled intended use. The investigator envisage that the endpoint of the study will be single operator intubation success rate.

DETAILED DESCRIPTION:
Despite the introduction of videolaryngoscopes, flexible bronchoscopic intubation (FBI), also known as fiberoptic intubation (FOI), remains a critical method for achieving tracheal intubation in patients with difficult airways. Unfortunately, however, FOI often requires two-operators for success. One operator is required to manipulate the flexible bronchoscope through the patient's upper airway and into their trachea, while the second operator applies one or more maneuvers (e.g., jaw thrust, anterior jaw lift, or lingual retraction) with or without the use of a commercially-available fiberoptic intubating airway.

Previous studies have demonstrated the effectiveness of the currently available FIAs, but also illustrate the frequent need for an assistant for successful FOI. In this study, an assistant performed a jaw lift and a chin lift in all subjects as well.

The air-Q and air-Q SP are commercially-available supraglottic airways (SGAs) that can be used for primary airway maintenance or as a conduit for FOI, as can be the Williams, Ovassapian, and Berman Intubating Airways. The air-Q products have the same overall geometrical design, but differ in their cuff inflating mechanisms, where the air-Q uses a traditional pilot balloon valve, while the air-Q SP utilizes a self-inflating cuff that dynamically adjusts according to the relative resistances to airflow between the patient's lungs and the device's cuff. In prior trials comparing the air-Q and air-Q SP with the two other commercially-available SGAs, the air-Q and air-Q SP bowl design provided a partial or full view of the vocal cords in 80-92% of subjects without requiring any additional airway maneuvers applied by an assistant (e.g., jaw thrust, anterior jaw lift, or lingual retraction) (Galgon, 2011; Galgon, 2015). Presumably, in these situations, successful tracheal intubation using the air-Q or air-Q SP could have been achieved by a single operator versus requiring one or more assistants. However, this potential performance advantage has not yet been tested. Therefore, the purpose of this study is to compare use of the air-Q SP against the WA for FBI performed by a single operator.

The air-Q SP, rather than the air-Q, is chosen for this study because its lack of a pilot balloon valve allows its stem to be easily shortened to ease device removal over the coaxially placed tracheal tube. The WA is chosen for this study because it has performed best in past trials and is the airway routinely used by the study principal investigator (PI) for FBI. Both devices are commercially-available and being used in the study in accordance with their labeled intended use.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years);
2. The patient is scheduled for an elective surgery or procedure that will take place in the UWHC main operating room, outpatient surgical center, or ambulatory procedure center; and
3. The patient's primary anesthesia care team has planned for general anesthesia with orotracheal intubation for airway maintenance.

Exclusion Criteria:

1. The patient is < 18 years of age;
2. The patient is non-English speaking;
3. The patient is known or believed to be pregnant;
4. The patient is a prisoner;
5. The patient has impaired decision-making capacity;
6. The patient is at increased risk for aspiration, including non-fasted or emergency surgery, and cases of uncontrolled gastroesophageal reflux disease, hiatal hernia, gastroparesis, esophageal dysmotility, prior esophagectomy, and/or emesis within twenty-four hours of the surgery or procedure;
7. The patient has limited mouth opening or oropharyngeal anatomy making successful placement of the study airway conduit unlikely;
8. The patient has airway exam features, a medical condition, or a past airway management history, which prompts the attending anesthesiologist to plan to maintain spontaneous ventilation during tracheal intubation;
9. The patient pre-operatively is requiring supplemental oxygen;
10. The patient has moderate to severe cardiac disease, as evidenced by a left ventricular ejection fraction of ≤ 50% on the most recent echocardiogram, severe aortic valve stenosis, atrial fibrillation with a resting pre-operative heart rate of ≥ 90 beats per minute, and/or known, multi-vessel coronary artery, managed conservatively with medical management or by intervention with multiple coronary artery stents or coronary bypass grafting; and
11. The patient has an allergy to glycopyrrolate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is single-operator intubation success. | 15 minutes
  The primary purpose of this study is to compare the single-operator intubation success using the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation.

SECONDARY OUTCOMES:
Time required for conduit placement | 15 minutes
  The secondary purposes of this study are to compare device performance characteristics and patient responses to use of the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation
Time required for each intubation attempt | 15 minutes
  The secondary purposes of this study are to compare device performance characteristics and patient responses to use of the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation
Overall intubation time | 15 minutes
  The secondary purposes of this study are to compare device performance characteristics and patient responses to use of the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation
Number of attempts required for conduit placement | 15 minutes
  The secondary purposes of this study are to compare device performance characteristics and patient responses to use of the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation
Number of attempts for successful intubation | 15 minutes
  The secondary purposes of this study are to compare device performance characteristics and patient responses to use of the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation
Number and types of assistive airway maneuvers (e.g., jaw thrust, lingual retraction, etc.) for successful intubation | 15 minutes
  The secondary purposes of this study are to compare device performance characteristics and patient responses to use of the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation
Successful intubation method | 15 minutes
  The secondary purposes of this study are to compare device performance characteristics and patient responses to use of the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation
Tracheal tube dislodgment rate during conduit removal | 15 minutes
  The secondary purposes of this study are to compare device performance characteristics and patient responses to use of the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation
Oxygen desaturation rate | 15 minutes
  The secondary purposes of this study are to compare device performance characteristics and patient responses to use of the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation
Post operative sore throat rate. | 4 hours
  The secondary purposes of this study are to compare device performance characteristics and patient responses to use of the air-Q SP versus the Williams Intubating Airway as a conduit for flexible bronchoscopic intubation

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Galgon, MD, MS, Principal Investigator — Department of Anesthesiology,University of Wisconsin, Madison, Wisconsin, United States, 53792
Locations (1):
- University of Wisconsin Hopital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Galgon RE, Schroeder KM, Han S, Andrei A, Joffe AM. The air-Q((R)) intubating laryngeal airway vs the LMA-ProSeal(TM) : a prospective, randomised trial of airway seal pressure. Anaesthesia. 2011 Dec;66(12):1093-100. doi: 10.1111/j.1365-2044.2011.06863.x. Epub 2011 Aug 22. PMID 21880031
- See also: Galgon RE, Schroeder KM, Han S, et al. The air-Q(®) intubating laryngeal airway vs the LMA-ProSeal(TM) : a prospective, randomised trial of airway seal pressure. Anaesthesia. 2011 Dec;66(12):1093-100. — https://www.ncbi.nlm.nih.gov/pubmed/21880031?dopt=Abstract